CLINICAL TRIAL: NCT02126280
Title: Cross-sectional Clinical Study of the Individual Profile of Activation of Circulating Blood Monocytes in Subjects With Preclinical Atherosclerosis.
Brief Title: Monocyte Activation in Preclinical Atherosclerosis
Acronym: MAPA
Status: Completed | Type: Observational
Sponsor: Institute for Atherosclerosis Research, Russia (Other)
Responsible Party: Sponsor
Other Study IDs: IAR-MAPA
Record Dates: First submitted 2014-04-23; First posted 2014-04-30 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: Atherosclerosis
Keywords: proinflammatory cytokines; anti-inflammatory cytokines; human monocytes; activation; biomarkers; asymptomatic atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Whole blood taken with anticoagulants for immediate monocyte isolation to be seeded in cell culture, and for preparation of plasma samples to be frozen for lipid analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Subclinical atherosclerosis: In vitro estimation of individual reactivity of monocytes in study participants with asymptomatic atherosclerotic plaques found in carotid arteries by ultrasound examination
  Interventions: Other: In vitro estimation of individual reactivity of monocytes
- Healthy subjects: In vitro estimation of individual reactivity of monocytes in study participants without ultrasound signs of subclinical carotid atherosclerosis
  Interventions: Other: In vitro estimation of individual reactivity of monocytes
- Diffuse intimal thickening: In vitro estimation of individual reactivity of monocytes in study participants with diffuse intima-media thickening of carotid arteries found at ultrasound examination
  Interventions: Other: In vitro estimation of individual reactivity of monocytes

INTERVENTIONS:
Other: In vitro estimation of individual reactivity of monocytes — Technique for isolation/separation of monocytes with culture purity more than 95 % CD14-positive cells according to flow cytometry, the share of viable cells at least 98% by trypan blue vital staining, capable of producing TNFa at concentration of at least 50 pg/ml when stimulated with 100 ng/ml IFN-gamma, and CCL18 at concentration at least 30 pg/ml when stimulated with 10 ng/ml interleukin.

SUMMARY:
The study of proinflammatory and anti-inflammatory cytokines and chemokines expression profiles in human monocytes to identify new effective biomarkers that have the best diagnostic potential in asymptomatic atherosclerosis.

DETAILED DESCRIPTION:
This project is the first step in creating a method for assessing an individual activity of macrophages. The problems addressed in the project are socially significant because of the high incidence of life-threatening diseases and their effects in the population. The method of evaluation of monocyte-macrophages activity in human blood will be based on the analysis of expression of cytokines and chemokines - markers of inflammatory and anti-inflammatory activity of macrophages. The most informative panel of cytokines and chemokines obtained during the project can be further used to create effective diagnostic tests.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged 40 to 74 years
* arterial normotension or mild arterial hypertension (systolic blood pressure <160 mm Hg, diastolic blood pressure <90 mm Hg)
* absence of chronic diseases demanding permanent drug administration (more than 2 month per year)

Exclusion Criteria:

* personal history of transient ischemic attacks
* personal history of chronic diseases demanding permanent drug administration (more than 2 month per year)
* personal history of life-threatening diseases
* indications for surgical treatment of atherosclerotic lesions localized in the extracranial brachiocephalic system

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The inclusion of healthy individuals, of apparently healthy persons with a predisposition to atherosclerosis, and subjects with subclinical atherosclerosis, according to the results of ultrasonographic examination of carotids, to achieve 80% statistical power (up to 50 study participants per group).
  Conducting experiments on obtaining the individual cultures of blood monocytes and stimulation of cells by proinflammatory and anti-inflammatory stimuli
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2012-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Development and optimization of the method of monocyte-macrophage isolation. | up to 1 years
  Technique for isolation/separation of monocytes with culture purity more than 95 % CD14-positive cells according to flow cytometry, the share of viable cells at least 98% by trypan blue vital staining, capable of producing TNFa at concentration of at least 50 pg/ml when stimulated with 100 ng/ml IFN-gamma, and CCL18 at concentration at least 30 pg/ml when stimulated with 10 ng/ml interleukin.

SECONDARY OUTCOMES:
Sample processing and parameter measurements. | up to 1 years
  Creating a collection of samples of the culture medium during cell stimulation into pro-inflammatory or anti-inflammatory phenotype.
  Definition of individual profiles of cell activation by the production of proinflammatory and anti-inflammatory cytokines and chemokines (C5a, IL-4, IL-32 alpha, CD40 ligand, IL-5, CXCL10, G-CSF, IL-6, CXCL11/I-TAC, GM-CSF , IL-8, CCL2, CXCL1, IL-10, MIF, CCL1, IL-12 p70, CCL3, ICAM-1, IL-13, CCL4, IFN-gamma, IL-16, CCL5, IL-1 alpha, IL -17, CXCL12, IL-1 beta, IL-17E, Serpin E1, IL-1ra, TNF-alpha, IL-2, IL-27, and TREM-1).
  Database generation on individual reactivity of monocytes-macrophages from healthy donors, individuals predisposed to atherosclerosis, and patients with asymptomatic atherosclerosis.
  Creating a collection of samples. Determination of concentrations of pro-inflammatory and anti-inflammatory markers.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander N Orekhov, PhD, DSc, Principal Investigator — Institute for Atherosclerosis Research
Locations (1):
- Institute for Atherosclerosis Research, Moscow, Russia

REFERENCES:
- [Background] Gratchev A, Ovsiy I, Manousaridis I, Riabov V, Orekhov A, Kzhyshkowska J. Novel monocyte biomarkers of atherogenic conditions. Curr Pharm Des. 2013;19(33):5859-64. doi: 10.2174/1381612811319330004. PMID 23438959
- [Background] Gratchev A, Sobenin I, Orekhov A, Kzhyshkowska J. Monocytes as a diagnostic marker of cardiovascular diseases. Immunobiology. 2012 May;217(5):476-82. doi: 10.1016/j.imbio.2012.01.008. Epub 2012 Jan 13. PMID 22325375